CLINICAL TRIAL: NCT06676306
Title: Patient and Caregiver Priorities in Neuro-Oncology Care
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-000229; NCI-2024-09052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000229 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Malignant Central Nervous System Neoplasm; Metastatic Malignant Neoplasm in the Central Nervous System
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational: Patients and their caregivers participate in interviews on study. Patients also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study is being done to identify patient and caregiver burdens regarding their experience with diagnosis and treatment of CNS tumors. These results will help doctors find areas where patients and caregivers may need more support.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe the patient experience and characterize the symptom burden related to primary or metastatic central nervous system tumors.

II. Describe the caregiver experience and caregiver needs related to patients with primary or metastatic central nervous system tumors. III. Establish which interventional treatment outcomes are important to patients and caregivers, within a wider understanding of their lived experience with CNS tumors and their treatment.

OUTLINE: This is an observational study.

Patients and their caregivers participate in interviews on study. Patients also have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Age ≥ 18 years.

  * Diagnosis of primary or metastatic CNS tumor with a primary caregiver, should patient wish to involve one.
  * Willing and able to participate in a semi-structured interview lasting approximately 60 minutes. Dyad interviews conducted for participants who elect to involve a caregiver.
  * Willing and able to participate in a single follow-up interview. Dyad follow up interviews conducted for participants who elect to involve a caregiver.

Exclusion Criteria:

* * Uncontrolled and/or intercurrent illness which limits participation in study interview.

  * Vulnerable populations: pregnant or nursing persons, prisoners, or persons lacking capacity for understanding.
  * Unable to read and speak English.

    * Note: English does not need to be primary language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of primary or metastatic CNS tumor with a primary caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient experience | Up to 6 months
  Participant and caregiver interviews will be analyzed qualitatively and reported descriptively. Interviews will be analyzed to describe the patient experience related to primary or metastatic central nervous system (CNS) tumors.
Symptom burden related to primary or metastatic central nervous system tumors | Up to 6 months
  Participant and caregiver interviews will be analyzed qualitatively and reported descriptively. Interviews will be analyzed to characterize the symptom burden related to primary or metastatic central nervous system (CNS) tumors.
Caregiver experience | Up to 6 months
  Patient and caregiver interviews will be analyzed qualitatively using thematic analysis and reported descriptively. Interviews will be analyzed to characterize the caregiver experience related to primary or metastatic CNS tumors.
Caregiver needs | Up to 6 months
  Patient and caregiver interviews will be analyzed qualitatively using thematic analysis and reported descriptively. Interviews will be analyzed to characterize caregiver needs related to primary or metastatic CNS tumors.
Importance of treatment outcomes | Up to 6 months
  Patient and caregiver interviews will be analyzed qualitatively using thematic analysis and reported descriptively. Interviews will be analyzed to establish which interventional treatment outcomes are important to patients and caregivers, within a wider understanding of their lived experience with CNS tumors and their treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ugur T. Sener, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials